CLINICAL TRIAL: NCT06040463
Title: Improving Diabetes Equity and Advancing Care Study
Acronym: IDEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinai Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 23-11
Record Dates: First submitted 2023-09-07; First posted 2023-09-15 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-09

CONDITIONS: Diabetes; Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: implementation science; optimization study
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART)
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Remote Glucose Monitoring > Remote Glucose Monitoring (RGM->RGM) (Experimental): Participant will be randomized into the RGM study arm for the first 6 months. At the 6-month rerandomization point, if the patient is a responder (A1c improved by at least 1 percentage point), patient will remain in the RGM group.
  Interventions: Behavioral: Remote Glucose Monitoring (RGM)
- Remote Glucose Monitoring > Remote Glucose Monitoring+Community Health Worker (RGM->RGM+CHW) (Experimental): Participant will be randomized into the RGM study arm for the first 6 months. At the 6-month rerandomization point, if the patient is a non-responder (A1c has not improved by at least 1 percentage point), patient will be randomized again with one arm being a continuation of RGM, with the addition of a CHW to provide tailored support.
  Interventions: Behavioral: Remote Glucose Monitoring (RGM); Behavioral: Community Health Worker tailored support
- Remote Glucose Monitoring > Diabetes Self-Management Training (RGM->DSMT) (Experimental): Participant will be randomized into the RGM study arm for the first 6 months. At the 6-month rerandomization point, if the patient is a non-responder (A1c has not improved by at least 1 percentage point), patient will be randomized again with one arm being diabetes self-management training (DSMT).
  Interventions: Behavioral: Diabetes Self-Management Training (DSMT); Behavioral: Remote Glucose Monitoring (RGM)
- Diabetes Self-Management Training > Standard of Care (DSMT->SOC) (Experimental): Participant will be randomized into the DSMT study arm for the first 6 months. At the 6-month rerandomization point, if the patient is a responder (A1c improved by at least 1 percentage point), patient will be directed back to standard of care.
  Interventions: Behavioral: Diabetes Self-Management Training (DSMT)
- Diabetes Self-Management Training > Community Health Worker (DSMT->CHW) (Experimental): Participant will be randomized into the DSMT study arm for the first 6 months. At the 6-month rerandomization point, if the patient is a non-responder (A1c has not improved by at least 1 percentage point), patient will be randomized again with one arm being a CHW to provide tailored support.
  Interventions: Behavioral: Diabetes Self-Management Training (DSMT); Behavioral: Community Health Worker tailored support
- Diabetes Self-Management Training > Remote Glucose Monitoring (DSMT->RGM) (Experimental): Participant will be randomized into the DSMT study arm for the first 6 months. At the 6-month rerandomization point, if the patient is a non-responder (A1c has not improved by at least 1 percentage point), patient will be randomized again with one arm being RGM.
  Interventions: Behavioral: Diabetes Self-Management Training (DSMT); Behavioral: Remote Glucose Monitoring (RGM)

INTERVENTIONS:
Behavioral: Diabetes Self-Management Training (DSMT) — The American Diabetes Association endorses the use of small-group diabetes self-management training (DSMT), for people living with diabetes to improve lifestyle, HbA1c levels, and overall quality of life. A certified diabetes care and education specialist will teach a four-part series of one-hour sessions providing culturally competent group education and discussion for groups of 5-8 patients: Session 1 - Living with diabetes - physiology of diabetes, integrating diabetes into your daily life, long term outcomes of diabetes; Session 2 - Culturally competent food education & portion control; Session 3 - Tips & Tricks for dining out and special occasions; Session 4 - Advanced tools and psychosocial implications of living with diabetes. While patients will be encouraged to move through the series together as a cohort, there will be make-up sessions and flexibility to ensure high-quality participation.
  Other Names: Diabetes Self-Management Education and Support (DSMES)
  Arms: Diabetes Self-Management Training > Community Health Worker (DSMT->CHW); Diabetes Self-Management Training > Remote Glucose Monitoring (DSMT->RGM); Diabetes Self-Management Training > Standard of Care (DSMT->SOC); Remote Glucose Monitoring > Diabetes Self-Management Training (RGM->DSMT)
Behavioral: Remote Glucose Monitoring (RGM) — Remote Glucose Monitoring (RGM) is an automated process of transmitting glucose levels directly from a personal smartphone device to a healthcare provider using a remote data transmitter. Since 2020, Sinai has worked with Glooko Inc. to provide the RGM platform and technical assistance to patients and for Sinai providers to access data remotely. Via the app, patients can: document their glucose levels; sync data from a meter, insulin pump, pen or continuous glucose monitoring device; track their weight; log food and meals; access educational resources; track steps; and track blood pressure. Remotely uploading data provides patients with a direct line to their provider for regular feedback on progress and answers to questions between clinic visits. Patients also receive one one-hour education session on RGM and the Glooko application.
  Arms: Diabetes Self-Management Training > Remote Glucose Monitoring (DSMT->RGM); Remote Glucose Monitoring > Diabetes Self-Management Training (RGM->DSMT); Remote Glucose Monitoring > Remote Glucose Monitoring (RGM->RGM); Remote Glucose Monitoring > Remote Glucose Monitoring+Community Health Worker (RGM->RGM+CHW)
Behavioral: Community Health Worker tailored support — CHWs are frontline public health workers who are trusted members of and/or have an unusually close understanding of the community served. The Center has two bilingual (Spanish/English) CHWs; additional bilingual CHWs will be added to the team to support the proposed study. While approaches will differ slightly depending on the patient and study condition, all patients paired with a CHW will be screened for social needs utilizing a standard social determinants of health (SDoH) screening tool, receive referrals to resources to address unmet social/health needs, and aided in navigating health and social systems.
  Arms: Diabetes Self-Management Training > Community Health Worker (DSMT->CHW); Remote Glucose Monitoring > Remote Glucose Monitoring+Community Health Worker (RGM->RGM+CHW)

SUMMARY:
The goal of this randomized trial is to determine the optimal combination and sequence of three enhancements for a team-based care model for patients living with diabetes in Chicago. The study aim is to determine optimization of intervention components. Participants will be randomly assigned to diabetes self-management training or remote glucose monitoring. After 6 months, participants will be rerandomized to a subsequent study arm (including a CHW support program) depending on a tailoring variable of change in A1c. Researchers will compare the final 6 study arms to see which combination and sequence of enhancements produces the most improvement in A1c.

DETAILED DESCRIPTION:
Sinai Health System is Illinois' largest private safety-net healthcare system, serving predominantly low-income communities of color with large Medicaid-eligible populations in Chicago. In response to high diabetes rates and community calls for coordinated, multidisciplinary diabetes care, Sinai designed the Center for Diabetes and Endocrinology (the Center) which launched in 2020. The Center uses a comprehensive model with streamlined services to address the full spectrum of patient medical and non-medical needs. This study seeks to determine the appropriateness and fidelity of three intervention components of a team-based care model for patients served by the Center to define the ideal sequence for improving patient outcomes. Grounded in qualitative methodology and guided by a sequential multiple assignment randomized trial (SMART), we propose evaluating the appropriateness of novel intervention components (Aim 1); measuring fidelity of new intervention components (Aim 2); comparing the effectiveness and determine optimization of intervention components (Aim 3). We will evaluate Aim 1 via key stakeholder interviews and focus groups. We will analyze Aims 2 & 3 by conducting descriptive statistics on all variables, giving special attention to outlier values. We will also run bivariate and multivariate analyses across variables of interest and time points to determine the optimal sequence of intervention activities.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 1 or type 2 diabetes
* 18+ years of age
* Able to provide consent
* Identify as African American/Black or Latinx
* most recent HbA1c > 7%,
* Have a smartphone compatible with the Glooko application
* Have completed at least one Center appointment (i.e. current patient)
* Completed at least 3 months of their assigned study condition

Exclusion Criteria:

* Already an active user of RGM
* Actively working with a CHW
* Diagnosis of gestational diabetes (without type 1 or type 2)
* Has a Power of Attorney
* Be suffering from Stage-V renal disease or undergoing dialysis.
* Be suffering from a severe form of cardiovascular disease (NYHA Class III and IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in A1c | Baseline (time = 0); 6 months (time = 1); 12 months (time = 2)
  Change in A1c from baseline to the 12-month study end point measured at the patient level. Measure will be collected every 6 months, at a minimum. The 6-month A1c will be used to determine their study condition at the rerandomization poiont.

SECONDARY OUTCOMES:
Active Usage of RGM | Data will be exported from the Glooko application monthly for the full 18 months of the trial period.
  Active usage will be defined as at least one upload of data within a 30-day period and at least 16 blood glucose entries within a 30-day period.
DSMT Attendance | Attendance data will be collected throughout the entire study period (18 months)
  We will collect # and proportion of attended DSMT classes by participant.
CHW Support Adherence | After rerandomization period (starting at 6 months post enrollment)
  Adherence to CHW engagement will include completing the initial education session with a CHW, competing a SDoH screener and at least three phone or in-person touchpoints over the 6-month intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Study protocol is currently available. Remaining information will be available upon study completion.

REFERENCES:
- [Derived] Jacobs J, Labellarte P, Margellos-Anast H, Garcia L, Qeadan F, Tingey B, Barnick K, Dougherty A, Wagener C. Improving Diabetes Equity and Advancing Care (IDEA) to optimize team-based care at a safety-net health system for Black and Latine patients living with diabetes: study protocol for a sequential, multiple assignment, randomized trial. Trials. 2024 Jul 24;25(1):504. doi: 10.1186/s13063-024-08346-9. PMID 39049044